CLINICAL TRIAL: NCT02729363
Title: The Feasibility of the PAINReportIt Guided Relaxation Intervention for Pain and Stress Symptoms in Adult Outpatients With Sickle Cell Disease
Brief Title: The Feasibility of the PAINReportIt Guided Relaxation Intervention-Outpatient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201600042
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Disease; Stress; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Relaxation video clip (Experimental): This intervention is a 12-minute guided audio-visual relaxation intervention delivered at the baseline visit to determine the immediate effects of guided relaxation intervention on stress and pain in outpatients with sickle cell disease.
  Interventions: Behavioral: Guided Relaxation video clip
- Sickle cell experience discussion (Other): Attention Control Group: This intervention is a 12-minute sickle cell disease experience discussion. In this computer-based discussion, patients talk about their sickle cell disease experience. The audio-taped questions and onscreen directions were programmed for self-administration. Subjects' responses will be captured via the microphone so that Data Collectors are not involved in this discussion process, and it is equivalent to the guided relaxation activity.
  Interventions: Behavioral: Sickle Cell Disease Experience Discussion

INTERVENTIONS:
Behavioral: Guided Relaxation video clip — This intervention is a 12-minute guided audio-visual relaxation intervention.
  Arms: Guided Relaxation video clip
Behavioral: Sickle Cell Disease Experience Discussion — This intervention is a 12-minute computer-administered sickle cell disease experience discussion.
  Arms: Sickle cell experience discussion

SUMMARY:
Our goal is to improve the self-management of pain and stress in adult outpatients with sickle cell disease (SCD) by determining the feasibility of a self-managed guided relaxation (GR) stress reduction intervention using a tablet-based mobile device. Currently, opioid analgesics are primarily used to treat SCD pain while self-managed behavioral modalities such as GR, are rarely used. Little is known about the effects or mechanisms of GR on pain and stress, in adults with SCD. Emerging evidence from the hypothalamic pituitary adrenal (HPA) axis theory offer insights for understanding the mechanisms. Adding GR as a supplement to analgesic therapies will address the paucity of self-management strategies for controlling pain in SCD. GR is a simple and cost-effective non-drug intervention that could reduce pain and stress in outpatients with SCD. GR is an intervention where outpatients with SCD are directed to listen to and view audio-visual recordings while they visualize themselves being immersed in that scene.

DETAILED DESCRIPTION:
The investigator will recruit adult outpatients with sickle cell disease (SCD) from the University of Florida Health Hematology Clinics and conduct study visits in a research room located at the College of nursing.

The investigator will stratify participants on worst pain intensity (<=5 and >5) and randomly assign 15 adults to attention control (stress/pain tracking; 12-min SCD experience discussion) and 15 adults to experimental (stress/pain tracking; 12-min GR video clip) groups.

The immediate intervention effects will be examined for pain (primary) and stress (secondary) outcomes. Vital signs for determining relaxation responses (mediators) will be collected immediately before and after the 12-min interventions.

ELIGIBILITY:
Inclusion Criteria:

* Has SCD diagnosis;
* Reports pain 3 or greater in the previous 24 hours (0-10 scale)
* Receives care at the University of Florida (UF) Health/Shands
* Speaks and reads English
* 18 years of age or older
* Self-identifies as being of African or Hispanic descent

Exclusion Criteria:

* Legally blind
* Physically or cognitively unable to complete study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02-23 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Current pain | Immediate (baseline)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain intensity scale: A 3-item scale that asks patients to report their pain now, worst, and average on a scale of 1 to 5 where 1 is "had no pain" and 5 is "very severe." We will estimate intervention effects using regression analysis.

SECONDARY OUTCOMES:
Current stress | Immediate (baseline)
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We will estimate intervention effects using linear regression.

OTHER OUTCOMES:
Physiologic markers of relaxation (pulse, respiration, finger temperature) | Immediate (baseline)
  Physiological markers of relaxation (pulse, respiration, finger temperature) will be measured using a standard vital sign measuring device. We will estimate intervention effects using regression analysis. We expect to observe trends for the immediate GR effect in terms of decreases in relaxation indicators (respiration rate, heart rate) and increases in skin temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam O Ezenwa, PhD, RN, Principal Investigator — University of Florida
Locations (1):
- University of Florida Hematology Clinic-Medical Plaza, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ezenwa MO, Yao Y, Nguyen MT, Mandernach MW, Hunter CT, Yoon SL, Fedele D, Lucero RJ, Lyon D, Wilkie DJ. Randomized Pilot Study: A Mobile Technology-based Self-management Intervention for Sickle Cell Pain. West J Nurs Res. 2020 Aug;42(8):629-639. doi: 10.1177/0193945919878821. Epub 2019 Oct 4. PMID 31583977